CLINICAL TRIAL: NCT03377166
Title: Measuring Subjective Visual Vertical (SVV) Using a Smartphone Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Director, Tel-Aviv Sourasky Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0113-17-TLV
Record Dates: First submitted 2017-12-07; First posted 2017-12-19 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Subjective Visual Vertical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vertigo (Active Comparator): Participants with vestibular disorder
  Interventions: Diagnostic Test: Bucket test and Smartphone-based evaluation of SVV
- Control (Active Comparator): Participants without vestibular disorder
  Interventions: Diagnostic Test: Bucket test and Smartphone-based evaluation of SVV

INTERVENTIONS:
Diagnostic Test: Bucket test and Smartphone-based evaluation of SVV — Bucket test and Smartphone-based evaluation of SVV

SUMMARY:
A comparison between two methods evaluating SVV: Bucket Test and A smartphone-based test.

ELIGIBILITY:
Inclusion Criteria:

* Vestibular Disorder

Exclusion Criteria:

* Chronic ear disease, Neurological disorder, s/p Ear surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Results of Bucket test Smartphone-based evaluation of SVV | 5 minutes
Results of Smartphone-based evaluation of SVV | 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- The Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No